CLINICAL TRIAL: NCT01878396
Title: Predictive Value of Circulating Melanoma Cells (CMCs) in Metastatic Melanoma (MM) Patients Treated With Selective Inhibitors of BRAF
Brief Title: Circulating Melanoma Cells in Metastatic Patients Treated With Selective BRAF Inhibitors
Acronym: CMCBRAF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Oncologico Veneto IRCCS (Other)
Collaborators: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: IOV2011/35; CE IOV 2011/35 (Other: Comitato Etico IOV)
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Metastatic Melanoma
Keywords: Circulating Melanoma cells in metastatic melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Mutated Anti-B-RAF: Fourth stage Melanoma patients with both measurable and not measurable lesions undergoing treatment with selective B-RAF inhibitors.
  Interventions: Drug: Anti-B-RAF

INTERVENTIONS:
Drug: Anti-B-RAF

SUMMARY:
The purpose of this study, is to evaluate Circulating Melanoma Cell (CMC) changes in Metastatic Melanoma (MM) patients, undergoing treatment with selective inhibitors of mutated BRAF.

DETAILED DESCRIPTION:
This is an observational prospective pilot study aimed to investigate the association between changes of total and apoptotic CMC count and disease progression in MM patients undergoing treatment with selective inhibitors of mutated B-RAF.

ELIGIBILITY:
Inclusion Criteria:

* Fourth stage Melanoma patients with both measurable and not measurable lesions undergoing treatment with selective B-RAF inhibitors will be included. To determine the prevalence of CMC-positive patients in IV stage Melanoma, patients without mutated B-RAF undergoing chemotherapy and/or vaccines will be also enrolled at baseline, as part of study protocols approved and activated in the participating centers.
* Informed written consent.

Exclusion Criteria:

* Inadequate compliance to multiple blood draws (baseline, 15 days, 1th month, 4th month, and/or at progression) as scheduled in this adjunctive biologic study for patients carrying B-FAF mutation; inadequate compliance to adjunctive blood draws, as scheduled at baseline for BRAF wild-type
* Previously exposure to immunological treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of CMC count during treatment and comparison with CT and PET | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paola Zanovello, Phd, Principal Investigator — Padua University
Locations (1):
- Vanna Chiarion-Sileni, MD, Padua, PD, Italy

REFERENCES:
- [Background] Rao C, Bui T, Connelly M, Doyle G, Karydis I, Middleton MR, Clack G, Malone M, Coumans FA, Terstappen LW. Circulating melanoma cells and survival in metastatic melanoma. Int J Oncol. 2011 Mar;38(3):755-60. doi: 10.3892/ijo.2011.896. Epub 2011 Jan 3. PMID 21206975
- [Background] Mocellin S, Hoon D, Ambrosi A, Nitti D, Rossi CR. The prognostic value of circulating tumor cells in patients with melanoma: a systematic review and meta-analysis. Clin Cancer Res. 2006 Aug 1;12(15):4605-13. doi: 10.1158/1078-0432.CCR-06-0823. PMID 16899608
- [Background] Rossi E, Basso U, Celadin R, Zilio F, Pucciarelli S, Aieta M, Barile C, Sava T, Bonciarelli G, Tumolo S, Ghiotto C, Magro C, Jirillo A, Indraccolo S, Amadori A, Zamarchi R. M30 neoepitope expression in epithelial cancer: quantification of apoptosis in circulating tumor cells by CellSearch analysis. Clin Cancer Res. 2010 Nov 1;16(21):5233-43. doi: 10.1158/1078-0432.CCR-10-1449. Epub 2010 Oct 26. PMID 20978147
- [Background] Rossi E, Fassan M, Aieta M, Zilio F, Celadin R, Borin M, Grassi A, Troiani L, Basso U, Barile C, Sava T, Lanza C, Miatello L, Jirillo A, Rugge M, Indraccolo S, Cristofanilli M, Amadori A, Zamarchi R. Dynamic changes of live/apoptotic circulating tumour cells as predictive marker of response to sunitinib in metastatic renal cancer. Br J Cancer. 2012 Oct 9;107(8):1286-94. doi: 10.1038/bjc.2012.388. Epub 2012 Sep 6. PMID 22955853
- [Background] Mocellin S, Del Fiore P, Guarnieri L, Scalerta R, Foletto M, Chiarion V, Pilati P, Nitti D, Lise M, Rossi CR. Molecular detection of circulating tumor cells is an independent prognostic factor in patients with high-risk cutaneous melanoma. Int J Cancer. 2004 Sep 20;111(5):741-5. doi: 10.1002/ijc.20347. PMID 15252844